CLINICAL TRIAL: NCT02319486
Title: CEV With/Without Periocular Carboplatin Chemotherapy for Nonmetastatic Extraocular Retinoblastoma Carboplatin--A Single Center, Retrospective Study to Evaluate the Efficacy of Carboplatin in Subjects With Retinoblastoma
Brief Title: CEV With/Without Periocular Carboplatin Chemotherapy for Extraocular Retinoblastoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Huasheng Yang, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yanghs04
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; carboplatin
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Vincristine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEV with/without carboplatin (Experimental): CEV chemotherapy(CEV Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months) together with/without 20mg/2ml carboplatin periocular injection
  Interventions: Drug: carboplatin periocular injection; Drug: CEV chemotherapy

INTERVENTIONS:
Drug: carboplatin periocular injection — chemotherapy together with/without 20mg/2ml carboplatin periocular injection
  Other Names: carboplatin
Drug: CEV chemotherapy — vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2
  Other Names: carboplatin,vincristine, etoposide

SUMMARY:
This study will evaluate a uniform chemotherapy protocol for nonmetastatic extraocular retinoblastoma

DETAILED DESCRIPTION:
This study will be a phase 4 open label interventional case series. Patients with retinoblastoma will be receive chemotherapy with or without periocular injections of carboplatin at a dose of 20mg/2 ml. Patients will receive chemotherapy on a monthly basis for a total duration of therapy of 6 months. Patients will be followed for 18 months .

ELIGIBILITY:
Inclusion Criteria:

* IRSS stage II or stage IIIa RB patients.
* for patients with IRSS stage II disease, if scleral surface invasion alone was observed, only systemic chemotherapy was administered, whereas other IRSS stage II and IIIa patients received systemic chemotherapy plus additional local chemotherapy.
* no tumor-related treatment was given prior to this chemotherapy regimen.

Exclusion Criteria:

* metastasis, including lymph node metastasis.
* the diagnosis of IRSS stage I or above in the non-target eye.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huasheng Yang, M.D, PHD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Object: Stage II or IIIa base on International Retinoblastoma Staging System dates: January 2009- February 2014 location: Zhongshan Ophthalmic Center
Pre-assignment Details: Exclusion Criteria:
  * Any previous disease in the study eye.
  * Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals).
  * History of chemical intervention for retinoblastoma in the study eye.
  * Over Stage I base on International Retinoblastoma Staging System for the other eye.
Period: Overall Study
Arm/Group | CEV With/Without Carboplatin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CEV With/Without Carboplatin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Full Range); unit: months] | 2.5 [1.5 to 7.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 21
Region of Enrollment [Number; unit: participants]
  China | 26
Number of Participants [Number; unit: participants]
  stage II | 9
  stage IIIa | 17

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Rate
Description: measure the event free survival rate for the patients at 18 months: patients that without tumor relapse or metastasis
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- CEV With/Without Carboplatin- Stage 2; CEV With/Without Carboplatin - Stage 3: CEV chemotherapy(CEV Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months) together with/without 20mg/2ml carboplatin periocular injection
  carboplatin periocular injection: chemotherapy together with/without 20mg/2ml carboplatin periocular injection
  CEV chemotherapy: vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2
Arm/Group | CEV With/Without Carboplatin- Stage 2 | CEV With/Without Carboplatin - Stage 3
Number analyzed (Participants) | 9 | 17
participants | 7 | 4
Statistical Analysis 1: Comparison: CEV With/Without Carboplatin- Stage 2 vs CEV With/Without Carboplatin - Stage 3; Test type: Superiority or Other; p = 0.034, pEFS — stage 2 vs stage 3; Probability of Event-Free Survival ，pEFS = 0.32 — over all pEFS

ADVERSE EVENTS:
Time Frame: up to 2 years
Groups:
- CEV With/Without Carboplatin-Stage 2; CEV With/Without Carboplatin-Stage 3: CEV chemotherapy(CEV Chemotherapy:vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2.monthly for the first six months) together with/without 20mg/2ml carboplatin periocular injection
  carboplatin periocular injection: chemotherapy together with/without 20mg/2ml carboplatin periocular injection
  CEV chemotherapy: vincristine,1.5mg/m2;carboplatin,560mg/ m2;etoposide,150 mg/ m2
Arm/Group | CEV With/Without Carboplatin-Stage 2 | CEV With/Without Carboplatin-Stage 3
Serious Adverse Events (participants affected / at risk) | 2/9 | 13/17
Other Adverse Events (participants affected / at risk) | 0/9 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CEV With/Without Carboplatin-Stage 2 (N=9) | CEV With/Without Carboplatin-Stage 3 (N=17)
central nervous system metastasis (Nervous system disorders) | 2 | 10
Orbit Relapse (Eye disorders) | 0 | 1
central nervous system metastasis and orbit relapse (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No